CLINICAL TRIAL: NCT05559736
Title: Pilot Evaluation: Artemis Proximal Femoral Nail (PFN) for Internal Fixation of Intertrochanteric Femur Fractures
Brief Title: Artemis Proximal Femoral Nail for Internal Fixation of Intertrochanteric Femur Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no interest in using implant
Sponsor: Johns Hopkins University (Other)
Collaborators: Innov8ortho (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00344949
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Intertrochanteric Fractures; Femoral Fracture; Femoral Neck Fractures
Keywords: Femoral nail; Cephalomedullary nail; Artemis Proximal Femoral Nail; Intertrochanteric femur fractures
MeSH Terms: conditions — Hip Fractures; Femoral Fractures; Femoral Neck Fractures | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Artemis Proximal Femoral Nail (PFN) implant (Experimental): All participants will receive the Artemis Proximal Femoral Nail (PFN) implant.
  Interventions: Device: Artemis Proximal Femoral Nail (PFN) implant

INTERVENTIONS:
Device: Artemis Proximal Femoral Nail (PFN) implant — Artemis Proximal Femoral Nail (PFN) implant

SUMMARY:
In February 2021, Altior Trauma Innovations™ announced that it had received 501(k) FDA approval for the Artemis Proximal Femoral Nail (PFN) System for internal fixation of intertrochanteric femur fractures. The objective of this pilot study is to evaluate safety, efficacy and feasibility of the Artemis PFN implant for operative fixation of intertrochanteric femoral fractures, compared to matched historical control patients who received other implants.

DETAILED DESCRIPTION:
Intertrochanteric femur fractures are a common injury pattern seen after acute hip trauma, with a very high rate of morbidity and mortality particularly among elderly patients. Cephalomedullary nail fixation has become a mainstay of treatment for both stable and unstable intertrochanteric fractures, offering greater stability than other options without replacing the native hip joint when possible. Despite this, the incidence of fracture nonunion remains high, resulting in poor functional outcomes, higher healthcare costs, and conversion to hemi- or total hip arthroplasty.

In February 2021, Altior Trauma Innovations™ announced that it had received 501(k) FDA approval for the Artemis Proximal Femoral Nail (PFN) System for internal fixation of intertrochanteric femur fractures. The Artemis PFN implant offers several purported advantages over existing implants. It is manufactured with a titanium core coated with carbon-fiber reinforced polyetheretherketone (PEEK), combining the strength of titanium with the bone-imitating biomechanical properties and radiolucency of PEEK. A number of additional features built into the Artemis System are designed to facilitate lower-complexity assembly/insertion, as well as reduce the likelihood of implant failure.

The objective of this pilot study is to evaluate safety, efficacy and feasibility of the Artemis PFN implant for operative fixation of intertrochanteric femoral fractures, compared to matched historical control patients who received other implants.

ELIGIBILITY:
Inclusion Criteria:

* All patients with traumatic, non-pathologic stable intertrochanteric fractures requiring cephalomedullary nail fixation

Exclusion Criteria:

* Pediatric patients (<18 years)
* Pregnant females
* Patients with other concomitant orthopaedic injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of fracture nonunion | Up to 6 months
Rate of implant-related failure | Up to 6 months

SECONDARY OUTCOMES:
Preoperative pain as assessed by a visual analog scale | 30 days preoperatively
  Visual Analog Scale: 1(least pain) - 10(most pain).
Preoperative function as assessed by the Functional Independence Measure | 30 days preoperatively
  Functional Independence Measure: 1(total functional dependence) - 7(total functional independence).
Operative duration | Intraoperative
  Operative duration in minutes.
Fluoroscopy usage time | Intraoperative
  Fluoroscopy usage time in minutes.
Estimated blood loss | Intraoperative
  Estimated blood loss in milliliters (mL).
Duration of hospital stay | Perioperative, up to 6 months post procedure
  Duration of hospital stay in days.
Discharge disposition | Perioperative, up to 6 months post procedure
  Discharge to home vs. rehab facility
Postoperative complications | Up to 6 months
  Any postoperative complications, including: infection, hematoma, thrombosis/embolism, delayed wound healing, etc.
Postoperative pain as assessed by a visual analog scale | Up to 6 months
  Visual Analog Scale: 1(least pain) - 10(most pain).
Postoperative function as assessed by the Functional Independence Measure | Up to 6 months
  Functional Independence Measure: 1(total functional dependence) - 7(total functional independence).
Use of gait-aid device | Up to 6 months
  Use of gait-aid device (wheelchair, walker, cane).
Postoperative radiographic healing | Up to 6 months
  Fracture healing, position of implant, implant-related failure (subsidence, cutout, loosening, implant fracture).
Financial costs | Intraoperative
  Implant purchase/manufacturing costs.
Environmental costs | Intraoperative
  Carbon waste footprint.

CONTACTS AND LOCATIONS:
Overall Officials: Amiethab Aiyer, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No